CLINICAL TRIAL: NCT02518906
Title: Process-Outcome Study on Psychotherapeutic Interventions in Adolescents With Personality Disorders
Brief Title: Evaluation of AIT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Schmeck (Other)
Collaborators: Heidelberg University (Other); Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor-Investigator, Klaus Schmeck, Professor of Child and Adolescent Psychiatry, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAST
Record Dates: First submitted 2015-07-16; First posted 2015-08-10 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Personality Disorders; Borderline Personality Disorder
Keywords: Psychotherapy; psychotherapy process; therapeutic alliance; psychotherapeutic change; psychophysiology
MeSH Terms: conditions — Personality Disorders; Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adolescent Identity Treatment (Experimental): Psychotherapeutic treatment performed routinely at the centres in Basel and Santiago de Chile
  Interventions: Behavioral: Adolescent Identity Treatment
- DBT-A (Experimental): Psychotherapeutic treatment performed routinely at the centre in Heidelberg
  Interventions: Behavioral: DBT-A

INTERVENTIONS:
Behavioral: Adolescent Identity Treatment — Integrative Approach for the treatment of adolescents with Personality Disorder.
  Manual was published in 2013.
  Arms: Adolescent Identity Treatment
Behavioral: DBT-A — Dialectic Behavioral Treatment for Adolescents is the most commonly used Approach for the Treatment of adolescents with Boderline Personality Disorder
  Arms: DBT-A

SUMMARY:
Specialized treatment of personality disorders (PD) in youth has been neglected for a long time, because these disorders were not diagnosed before the age of 18. Since 2013 the age threshold has been dropped in the Diagnostic and Statistical Manual (DSM)-5, and such change is also announced for the International Classification of Diseases (ICD)-11. There is broad consensus from both scientific evidence and clinical experience that specialized early interventions in adolescents with PD are urgently needed.

In the last decades a number of specialized psychotherapeutic treatment programs have been developed. Despite their conceptual differences, many of the treatment models have shown significant effects in the treatment of PD in adults. However, the treatment of adolescents with PD remains difficult and further enhancement and development of treatments is needed.

Given the different therapeutic approaches available, the present project aims to go beyond the comparison of integral therapeutic models in the classical outcome study design. While outcome research is important to build on the evidence of the effectiveness of an intervention, it contributes little to its understanding and refinement. The aim of the present multi-center project is to compare two therapeutic methods used in routine care:

* Adolescent Identity Treatment (AIT)
* Dialectic Behavioral Treatment for Adolescents (DBT-A)

Treatments will be performed at different study centers and compared using the same measures of outcome. The main outcome will be psychosocial functioning.

Additionally, the psychotherapy process will be investigated to explore specific and unspecific mechanisms of the therapeutic process, its outcome and mediators.

ELIGIBILITY:
Inclusion Criteria:

* Identity Diffusion (AIDA T-score > 60)
* borderline Criteria (SKID-II)

Exclusion Criteria:

* intelligence quotient (IQ) < 80
* psychotic disorder
* pervasive developmental disorders
* heavy and persistent substance abuse
* major somatic or neurological disease
* hospital treatment

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change in Children's Global Assessment Scale (CGAS) | Baseline, 12 months after Baseline
  Psychosocial functioning. Rated considering the results of the Columbia Impairment Scale - parent and patient versions

SECONDARY OUTCOMES:
Psychosocial functioning | Baseline, 12 months after Baseline
  Columbia Impairment Scale (CIS) (Patient and Parent versions)
School functioning | Baseline, 12 months after Baseline
  School Functioning Rating (SFR)
Change in Psychopathology | Baseline, 12 months after Baseline (only Basel and Heidelberg)
  Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID)
Change in Severity of Psychopathology | Baseline, 12 months after Baseline
  Clinical Global Impression Scale
Change in Depression | Baseline, 12 months after Baseline
  Beck Depression Inventory (BDI)
Change in Psychopathological Symptoms | Baseline, 12 months after Baseline
  Strengths & Difficulties Questionnaires (SDQ)
Change in Personality Functioning | Baseline, 12 months after Baseline (only Basel and Heidelberg)
  Levels of Personality Functioning - Questionnaire for Adolescents (LoPF-QA)
Change in Identity | Baseline, 12 months after Baseline
  Assessment of Identity Development in Adolescence (AIDA)
Change in Personality Disorder Symptoms | Baseline, 12 months after Baseline (only Basel and Heidelberg)
  Structured Clinical Interview of Diagnostic and Statistical Manual of Mental Disorders (DSM) (SCID)-II
Change in Interpersonal Problems | Baseline, 12 months after Baseline (only Santiago)
  Inventory of Interpersonal Problems (IIP-64)
Change in Mentalizing Capacity | Baseline, 12 months after Baseline
  Movie for the Assessment of Social Cognition (MASC)
Change in Quality of Life | Baseline, 12 months after Baseline
  Health-related Quality of Life Screening Instrument for Children and Adolescents (KIDSCREEN)
Change in Parental Stress | Baseline, 12 months after Baseline (only Basel and Heidelberg)
  Eltern-Belastungs-Inventar (EBI)
Self-injurious Behavior | Baseline, 12 months after Baseline (only Basel and Heidelberg)
  Self- Injurious Thoughts and Behaviors Interview
Borderline-specific Personality Pathology | Baseline, 12 months after Baseline (only Basel and Heidelberg)
  Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD)
Borderline-specific Symptoms | Baseline, 12 months after Baseline (only Basel and Santiago)
  Borderline Symptom List 23 (BSL-23)
Change in Psychophysiological Measures (Only Basel and Heidelberg) | Baseline, 12 months after Baseline
  Regression analysis will be used to evaluate change; Parameters: Heart Rate Variability and Electrodermal Activity (Basel only)
Change in Hair Cortisol Level (only Basel and Heidelberg) | Baseline, 12 months after Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schmeck, Prof., Study Director — University Basel
Locations (3):
- Millennium Institute for Research in Depression and Personality - Pontificia Universidad Católica de Chile, Santiago, Chile
- Department of Child and Adolescent Psychiatry, Centre for Psychosocial Medicine, University of Heidelberg, Heidelberg, Germany
- Psychiatric Universitiy Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmeck K, Weise S, Schluter-Muller S, Birkholzer M, Furer L, Koenig J, Krause M, Lerch S, Schenk N, Valdes N, Zimmermann R, Kaess M. Effectiveness of adolescent identity treatment (AIT) versus DBT-a for the treatment of adolescent borderline personality disorder. Personal Disord. 2023 Mar;14(2):148-160. doi: 10.1037/per0000572. Epub 2022 May 19. PMID 35587408
- [Derived] Zimmermann R, Furer L, Schenk N, Koenig J, Roth V, Schluter-Muller S, Kaess M, Schmeck K. Silence in the psychotherapy of adolescents with borderline personality pathology. Personal Disord. 2021 Mar;12(2):160-170. doi: 10.1037/per0000402. Epub 2020 Apr 23. PMID 32324008